**Title:** A RCT Evaluating Efficacy of Type-I Collagen Skin Substitute vs. Human Amnion Membrane in Treatment of Venous Leg Ulcers

**NCT No:** NCT06831760

**Date:** July 8, 2025

## **Study Aims**

This randomized, controlled clinical trial aimed to compare clinical efficacy, healing outcomes, of High Purity Type-I Collagen Skin Substitute (HPTC) vs. Dehydrated Human Amnion / Chorion Membrane (dHACM) in the treatment of venous leg ulcers.

## **Sample Size Calculation**

## Standard Two-Sample Comparison of Proportions (e.g., wound closure rate)

Assuming:

- $\alpha = 0.05 (5\%)$
- **Power** = 0.80 (80%)
- Proportion of success in control  $(p_1) = 0.60$  (typical healing rate for dHACM)
- **Proportion of success in treatment (p<sub>2</sub>)** = 0.90 (expected improvement with Type-I collagen)

We use the formula for comparing two proportions:

$$n=(p1-p2)2(Z\alpha/2+Z\beta)2\cdot[p1(1-p1)+p2(1-p2)]$$

Where:

- $Z\alpha/2Z_{\alpha/2} = 1.96$  for  $\alpha = 0.05$
- $Z\beta Z \{ beta \} Z\beta = 0.84 \text{ for } 80\% \text{ power}$

 $n = (1.96 + 0.84) 2 \cdot [0.6(0.4) + 0.9(0.1)](0.9 - 0.6) 2 = 7.84 \cdot [0.24 + 0.09]0.09 = 7.84 \cdot 0.330.09 = 2.590.09$   $\approx 28.8n$ 

We use the formula for comparing two proportions:

$$n = rac{(Z_{lpha/2} + Z_eta)^2 \cdot [p_1(1-p_1) + p_2(1-p_2)]}{(p_1 - p_2)^2}$$

Where:

- $Z_{\alpha/2}$  = 1.96 for  $\alpha$  = 0.05
- $Z_{eta}$  = 0.84 for 80% power

$$n = \frac{(1.96 + 0.84)^2 \cdot [0.6(0.4) + 0.9(0.1)]}{(0.9 - 0.6)^2} = \frac{7.84 \cdot [0.24 + 0.09]}{0.09} = \frac{7.84 \cdot 0.33}{0.09} = \frac{2.59}{0.09} \approx 28.8$$

 $\sim$ 29 participants per group - 30 per group is statistically adequate to detect a difference from 60% to 90% healing rate with 80% power.

**Randomization and Blinding:** Patients were randomized 1:1 to the HPTC or dHCAM group using a computer-generated randomization sequence. Open-label design (patients and clinicians were aware of treatment allocation). Outcome assessors and statisticians were blinded.

## **Data Collection and Monitoring**

- a. Baseline data: Demographics, medical history, ulcer characteristics.
- b. Weekly follow-ups: Wound measurements (photographic documentation), assess healing progress, pain scores, record adverse events and patient-reported outcomes.
- c. Histopathological specimens were obtained at baseline and day 5 for vascularity assessment.
- d. End-of-Study Visit (Week 6): final wound assessment, collect patient feedback on treatment experience, quality of life and scar assessment.
- e. Data entry and monitoring was managed using an electronic data capture system.

**Data Analysis:** Data was analysed using SPSS v26.0. Continuous variables were expressed as mean± standard deviation, and categorical variables as frequencies and percentages. Student's t-test was used for comparing continuous variables between groups, and chi-square test for categorical variables. A p-value <0.05 was considered statistically significant. Kaplan-Meier survival analysis was used to assess time to complete healing and Cohen's d values for primary histopathological parameters.